CLINICAL TRIAL: NCT03801031
Title: Sexual Dysfunction in Gynecologic Oncology Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: David Bender (Other)
Responsible Party: Sponsor-Investigator, David Bender, Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 201609770
Record Dates: First submitted 2019-01-09; First posted 2019-01-11 (Actual); Results first posted 2022-12-06 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-11

CONDITIONS: Gynecologic Cancer; Sexual Dysfunction
MeSH Terms: conditions — Sexual Dysfunction, Physiological | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lidocaine (Active Comparator): Patients being treated for gynecologic cancer assigned aqueous lidocaine solution as intervention to use during sexual encounters.
  Interventions: Drug: Lidocaine Topical
- Placebo (Placebo Comparator): Patients being treated for gynecologic cancer assigned placebo solution as intervention to use during sexual encounters.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lidocaine Topical — Many women treated for gynecologic cancer complain of sexual dysfunction and discomfort. It is thought that topical lidocaine application prior to sexual encounters may have reduced discomfort and improved overall quality of life during and following cancer treatment. The use of the lidocaine solution/placebo is the intervention.
  Arms: Lidocaine
Drug: Placebo — Placebo solution intervention used to validate the effects of the lidocaine solution usage.
  Arms: Placebo

SUMMARY:
This project will evaluate sexual dysfunction in women who have had surgery for gynecologic cancer. The subjects will complete a set of questionnaires about health, daily living, sexual encounters, and pain before their surgery and three times following. Each subject will be randomized to receive either lidocaine or a placebo that is applied vaginally immediately prior to any sexual encounters for approximately 6 months while maintaining a journal of sexual encounters and pain. The subjects and healthcare providers will be blinded to the treatment randomization until intervention and data collection is complete. Total participation will last up to one year from the date of enrollment. Subjects will visit the clinic at the same time as regular cancer care visits, receive the blinded intervention and complete the surveys.

DETAILED DESCRIPTION:
Once consented, subjects will complete nine short surveys (The Female Sexual Function Index, The PHQ-9, the GAD-7, the Social Provision Score (SPS), Rosenberg's Body Self-Esteem Index, the Severity of Posttraumatic Stress (PTS) Symptoms Scale, the Adverse Childhood Events Index, the Short Form (SF)-12, and the Dyadic Adjustment Scale) at their initial visit, assessing physical, psychological, and social elements related to sexuality.

Subjects will then have the tumor reduction surgery.

Twelve weeks after her surgery, each subject will be asked to complete the same nine-survey packet.

Once the second packet is completed, subjects will be randomized to receive either aqueous lidocaine (4%) or placebo with instructions to apply the solution to three cotton balls and place them on the perineum/vaginal introitus for one minute prior to sexual intercourse. Subjects will be educated on the use of this blinded intervention and be asked to keep a diary of sexual encounters, including a simple pictorial pain scale for each encounter. Subjects and providers are blinded to the assigned intervention.

Once subjects complete three months of perineal intervention, they will be asked at a follow-up visit (12 weeks following randomization) to complete the survey packet for a third time.

Subjects will then continue their perineal intervention, keep a diary of sexual encounters with the pain scale and return after another three-month interval for a fourth completion of the survey packet. Sexual encounter diaries and pain scale assessments will be collected and their participation in the trial will conclude. Also at the time of this concluding follow-up visit in the Gynecologic Oncology Clinic, patients will receive counseling by a gynecologic oncologist regarding education about sexual dysfunction, the possibility of experiencing sexual dysfunction, and a potential referral for further treatment of sexual dysfunction. The subject will remain blinded to the randomized intervention until the conclusion of the study.

Subjects will be unblinded and informed of assigned intervention at the conclusion of the study via a letter sent to their home address from the researchers.

ELIGIBILITY:
Inclusion criteria

* Female
* Age 18-99
* Planned to undergo primary surgical treatment at the University of Iowa Hospitals and Clinics for a suspected or proven diagnosis of ovarian, fallopian tube, peritoneal, endometrial, or cervical cancer
* Able to give informed consent and follow study procedures
* No previous reactions to lidocaine applications
* Performance Status of 0 or 1
* Reports having engaged in vaginal intercourse at least once in the last 12 months

Exclusion criteria:

* Failure to confirm invasive ovarian, fallopian tube, peritoneal, endometrial or cervical cancer by pathology from primary biopsy or surgery (subjects will not be eligible to continue the trial beyond the initial completion of the questionnaires)
* Diagnosis of another malignancy within the past five years, excluding basal cell carcinoma of the skin
* Patients undergoing primary or adjuvant external pelvic radiation (excluding adjuvant vaginal brachytherapy)
* Previous reactions to lidocaine applications
* Previous reactions to lidocaine for the subjects' sexual partner(s)

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2021-11-03 (Actual); Study Completion 2021-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Bender, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abbott-Anderson K, Kwekkeboom KL. A systematic review of sexual concerns reported by gynecological cancer survivors. Gynecol Oncol. 2012 Mar;124(3):477-89. doi: 10.1016/j.ygyno.2011.11.030. Epub 2011 Nov 28. PMID 22134375

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects will complete nine short surveys at their initial visit, assessing physical, psychological, and social elements related to sexuality. Subjects will then have the tumor reduction surgery. Twelve weeks after surgery, each subject will be asked to complete the same nine-survey packet. Once the second packet is completed, subjects will be randomized to receive either the lidocaine solution or a placebo using permuted block technique based on cancer origin.
Period: Overall Study
Arm/Group | Lidocaine | Placebo
Started | 3 | 1
Completed | 1 | 0
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Unable to comply | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lidocaine | Placebo | Total
Number analyzed (Participants) | 3 | 1 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Full Range); unit: years] | 56 [41 to 68] | 52 [52 to 52] | 55 [41 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Changes in Sexual Function
Description: Sexual function measured by the Female Sexual Function Index (FSFI) survey, a 19-item self-report survey measuring sexual function. Item responses are on a 5-point scale and the total scores range 2 to 36 points, considering that the higher the score obtained, the better the sexual function of the woman.
Time Frame: 9 months
Population: Study terminated prior to completion. Data not collected. Enrollment was halted prematurely and will not resume. Participants are no longer being examined or treated.
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Changes in Pain
Description: Pain is measured by using the visual analog scale for pain, which is a scale of 0-10, utilizing numbers and face illustrations to describe pain level. Pain level is measured on a 0-10 point scale, 0 indicating no pain and 10 indicating the worst pain possible.
Time Frame: 9 months
Population: as for outcome 1
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Depressive Symptoms
Description: Mean Change in Patient Health Questionnaire 9 (PHQ-9), a 9-item self-report instrument to screen for depression. Responses range from 0-3 and the scores range from 0-27, the higher total score indicates more depression.
Time Frame: 9 months
Population: as for outcome 1
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Anxiety
Description: Mean change in Generalized Anxiety Disorder 7-item scale (GAD-7), a brief self-report instrument of 7 items to assess generalized anxiety disorder. Responses range from 0-3 and the scores range from 0-21, the higher total score indicates more anxiety.
Time Frame: 9 months
Population: as for outcome 1
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Relationships and Social Support
Description: Mean change in Social Provisions Scale, a 24-item self-reported survey measuring perceived social support to assess confounders on sexual function. Responses range from 1-4 and higher total scores indicate greater social connection.
Time Frame: 9 months
Population: as for outcome 1
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Self-Esteem
Description: Mean change of Rosenberg's Body Self-Esteem Index, a 10-item self-report survey assessing global self-worth by measuring both positive and negative feelings about the self. Total scores range between 0 and 40; higher scores indicate better self-esteem.
Time Frame: 9 months
Population: as for outcome 1
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Posttraumatic Stress Symptoms
Description: Scores of Severity of Posttraumatic Stress Symptoms-Adult survey, a 9-item self-report instrument that assesses severity of posttraumatic stress disorder following a particular event or experience. Responses range from 0-4, 0 indicating no distress and 4 indicating extreme distress. Each item is measured on a 5-point scale (0=not at all; 4=extremely). Total score can range from 0-36 or averaged for 0-5. The higher scores indicate more severe PTS distress.
Time Frame: 9 months
Population: as for outcome 1
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Adverse Childhood Events
Description: Presence, Severity, or Mean Change in Adverse Childhood Events Index, a 10-item self-report scale measuring types of physical, verbal, and emotional childhood trauma. Items are responded with yes or no. The total score is the sum of yes responses and range from 0-10. Higher total scores indicate more adverse childhood experiences.
Time Frame: 9 months
Population: as for outcome 1
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Health Status
Description: Mean Change in SF-12, a 12-item self-report measure of perceived general health status and disability. Responses include yes or no or ranges on 5- or 6-point scales. Higher total scores indicate more disability.
Time Frame: 9 months
Population: as for outcome 1
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Romantic Relationships
Description: Mean Change in Dyadic Adjustment Scale (DAS), a 32-item self-report measure of couple satisfaction. Responses are 5- or 6-point scales or yes or no. Total scores range from 0 to 151. Higher total scores indicate higher adjustment and satisfaction in intimate relationships.
Time Frame: 9 months
Population: as for outcome 1
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Study participants will be asked if there have been any reactions to the solution supplied for perineal application at each clinic visit, up 6 months post-surgical intervention.
Arm/Group | Lidocaine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/1
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/1
Other Adverse Events (participants affected / at risk) | 0/3 | 0/1

LIMITATIONS AND CAVEATS:
This study stopped accrual early due to unmet targeted accrual goals with 4 subjects accrued out of 120 planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-02): https://cdn.clinicaltrials.gov/large-docs/31/NCT03801031/Prot_SAP_000.pdf
  • Informed Consent Form (2019-05-29): https://cdn.clinicaltrials.gov/large-docs/31/NCT03801031/ICF_001.pdf